CLINICAL TRIAL: NCT06640998
Title: Clinical Study to Evaluate the Safety and Efficacy of Matrix Pro Applicator Treatment to Lift the Eyebrow and Lift Lax Tissue in the Submentum and Neck
Brief Title: Safety and Efficacy of Matrix Pro for Eyebrow Lift and Lift of Submental/Neck Laxity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MXP24001
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Laxity; Skin
Keywords: Laxity; Brow Lift; Neck Lift; Sagging; Skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Zone 1: Eyebrow Lift (Experimental): Treatment of the upper face including treatment of forehead to mid cheek
  Interventions: Device: Matrix Pro
- Zone 2: Submentum and Neck (Experimental): Treatment of the lower face including mid to low cheek, submentum, and neck
  Interventions: Device: Matrix Pro

INTERVENTIONS:
Device: Matrix Pro — Study subjects received up to three (3) study treatments with the Matrix Pro applicator

SUMMARY:
Prospective, non-randomized, multi-center, pivotal clinical trial

DETAILED DESCRIPTION:
This is a two-arm study. Eligible participants will receive up to three treatments with the Matrix Pro Applicator for lifting the eyebrow and/or improving lax tissue in the submental and neck areas. Treatments will be spaced approximately 6 weeks apart (± 2 weeks), and all participants will undergo follow-up evaluations at 1 month (± 2 weeks) and 3 months (± 2 weeks) after the final treatment.

Each investigational site will treat two areas: In arm 1, the upper face, including the forehead and peri-orbital area, to lift the eyebrows. In arm 2, the lower face, including the submental and neck areas, to lift lax tissue. Each patient could be assigned to both arms. Treatment may occur immediately after the screening and enrollment visit or at a later date, depending on site scheduling. Additional follow-up visits may be required at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 75 years of age with Fitzpatrick Skin Type I - VI.
2. Presence of laxity to the eyebrow and/or submentum and neck appropriate for RF microneedling treatment.
3. Willing to receive Matrix treatments with The Matrix Pro applicator.
4. Able and willing to comply with the treatment/follow-up schedule and with all study (protocol) requirements.
5. Willingness to provide signed, informed consent to participate in the study.
6. Willing to abstain from neuromodulators, injectable fillers and any aesthetic procedure which may resurface the skin and/or modify the dermal tissue throughout the entire study duration.
7. Willing to abstain from other aesthetic procedures which may change or modify the eyelashes and/or eyebrows throughout the entire study duration.
8. Willing to maintain stable weight and avoid fluctuations of +/- 8lbs throughout the entire study duration.
9. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications, presentations, and marketing materials.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3-months prior to enrollment into the study, and/or breast feeding.
2. Pacemaker, internal defibrillator, or any active electrical implant anywhere in the body.
3. Superficial metal or other implants in the treatment area, unless these implants can be removed or covered with rolled gauze during treatment, except superficial dental implants.
4. Severe eyebrow heaviness/Laxity and/or severe submental fullness/ laxity of neck skin.
5. Weight has fluctuated +/- 8lbs within the past year.
6. Skin cancer in the treatment area or history of melanoma.
7. History of or current cancer and/or subject has undergone chemotherapy within the last 12 months.
8. Severe concurrent conditions, such as uncontrolled cardiac disorders, or poorly controlled endocrine disorders (diabetes or Hyper/Hypothyroidism).
9. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
10. Herpes Simplex Virus (HSV) in the intended treatment area unless treated following initiation of a prophylactic regimen.
11. Active skin condition in the treatment area such as sores, psoriasis, eczema, or rash, open wounds, and/or severe active inflammatory acne.
12. History of abnormal wound healing, keloid, or hypertrophic scar formation.
13. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitis disorders.
14. Known allergy to medication to be used during treatments such as lidocaine, benzocaine, tetracaine, Xylocaine, or Pro-Nox™ (a 50% oxygen and 50% nitrous oxide mixture (laughing gas).
15. On systemic corticosteroid therapy in past six months.
16. Currently taking anticoagulants.
17. Tattoos in the intended treatment area
18. Excessively tanned skin.
19. Is unwilling to have hair shaved from the treatment area, if applicable.
20. Facelift and/or neck lift in the last 12 months.
21. Aesthetics treatments/procedures (e.g. facial resurfacing and deep chemical peeling) within the last 4 months within the intended treatment area.
22. Neuromodulator injections (e.g. Botox®), collagen, non-permanent soft-tissue and/or dermal filler, and/or fat injections or other methods of augmentation with injected biomaterial in the treated area within the last 6-months.
23. Permanent synthetic fillers (e.g. silicone) or non-absorbable threads in the treatment area.
24. Absorbable facial threads within the last 2 years.
25. In the opinion of the Investigator, the subject is unwilling or unable to adhere to the study requirements or is otherwise unsuitable for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Improvements in lifting of lax tissue | 3 months post last treatment
  as assessed by independent masked evaluators of pre and post treatment images

CONTACTS AND LOCATIONS:
Locations (1):
- Candela Institute for Excellence, Marlborough, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No